CLINICAL TRIAL: NCT07330934
Title: A Multi-Center, Randomized, Double-Blind, Parallel, Placebo-Controlled Phase 2 Study to Evaluate the Efficacy and Safety of IBI356 in Adult Participants With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate Efficacy and Safety of IBI356 in Participants With Moderate to Severe Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI356A201
Record Dates: First submitted 2025-12-15; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- IBI356 dose 4 (Experimental): Participants receive IBI356 through W16
  Interventions: Drug: IBI356
- IBI356 dose 2 (Experimental): Participants receive IBI356 through W16
  Interventions: Drug: IBI356
- Dupilumab (Experimental): Participants receive dupilumab through W16
  Interventions: Drug: Dupilumab
- IBI356 dose 5 (Experimental): Participants receive IBI356 through W16
  Interventions: Drug: IBI356
- IBI356 dose 1 (Experimental): Participants receive IBI356 through W16
  Interventions: Drug: IBI356
- Placebo (Placebo Comparator): Participants receive placebo through W16
  Interventions: Drug: Placebo
- IBI356 dose 3 (Experimental): Participants receive IBI356 through W16
  Interventions: Drug: IBI356

INTERVENTIONS:
Drug: Dupilumab — Dupilumab by subcutaneous injection
  Arms: Dupilumab
Drug: Placebo — Placebo by subcutaneous injection
  Arms: Placebo
Drug: IBI356 — IBI356 by subcutaneous injection
  Arms: IBI356 dose 1; IBI356 dose 2; IBI356 dose 3; IBI356 dose 4; IBI356 dose 5

SUMMARY:
This is a multi-center, randomized, double-blind, parallel, placebo-controlled phase 2 clinical study. A total of 403 adult participants with moderate to severe AD are planned to be enrolled to evaluate efficacy, safety, PK characteristics, immunogenicity, and changes in PD characteristics of IBI356.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and sign the informed consent form (ICF);
2. Aged ≥ 18 years, male or female;
3. Diagnosis of AD for at least 1 year (defined by the American Academy of Dermatology Consensus Criteria);
4. EASI score of 16 or higher at baseline, vIGA-AD of 3 or 4 at baseline, AD involvement of 10% or more of BSA at baseline, weekly average of daily PP-NRS of ≥ 4 at baseline;
5. Participants with documented inadequate response to topical medications or for whom topical treatments are otherwise medically inadvisable.

Exclusion Criteria:

1. Presence of diseases that may affect the safety or efficacy, including but not limited to psychistric disorders, central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, and hematological or metabolic system diseases.
2. Known history of active tuberculosis or clinically suspected tuberculosis; or chest imaging suggesting evidence of suspected tuberculosis; or any other clinical evidence of latent tuberculosis.
3. Has known or suspected helminth or other parasitic infection.
4. History of malignancy, except excised or curatively treated localized basal cell carcinoma (BCC) or cutaneous squamous cell carcinoma (cSCC).
5. History of severe drug allergy or anaphylaxis.
6. Fainting, hemophobia, or inability to tolerate venipuncture.
7. Women who are pregnant or breastfeeding, or female participants who have a positive pregnancy test at screening or randomization.
8. Have received an organ or hematopoietic stem cell transplant.
9. Positive HBsAg; or positive HBcAb with positive HBV-DNA; or positive hepatitis C antibody with positive HCV-RNA; or positive treponema pallidum antibody; or positive HIV serology at screening.
10. Having received any of the specified therapy within the specified timeframe(s) prior to the baseline visit.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in Eczema Area and Severity Index (EASI) score | week 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.

SECONDARY OUTCOMES:
Proportion of participants achieving Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) of 0 (clear) or 1 (almost clear) with a ≥2-point reduction | week 16, 24
  The vIGA-AD is sn investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Proportion of participants with EASI-75/90/100 | week16, 24
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Proportion of participants with a ≥4-point reduction from baseline in the weekly average of the Peak Pruritus-Numerical Rating Scale (PP-NRS) | week 16, 24
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Change in EASI from baseline | Baseline to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Change in DLQI from baseline | Baseline to Week 48
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Change in POEM from baseline | Baseline to Week 48
  The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms on a 5-point scale; 0 (no days) to 4 (every day in the last week). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (very severe). Higher scores indicated more severe disease and poor quality of life.
Incidences of adverse events (AEs), treatment emergent adverse events (TEAEs), and serious adverse events (SAEs) | Baseline to Week 48
Serum IBI356 concentrations at prespecified timepoints | Baseline to Week 24
Percentage of Participants with Treatment-emergent ADA of IBI356 | Baseline to Week 24
Serum IL-13 (PD marker) be assessed as dose-dependent drug responses | Baseline to Week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China